CLINICAL TRIAL: NCT05610319
Title: Treat & Extend Versus Fixed Dosing with Faricimab for Management of Diabetic Macular Edema: a Pragmatic, Multi-center, Open-label, Randomized, Controlled Trial
Acronym: INSITE-DME
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-01; MR44143 (Other: Roche)
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Macular Edema
Keywords: Treat and Extend; Faricimab; Anti-VEGF
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Intervention Model Description: Two-armed, parallel, non-inferiority randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treat and Extend (Experimental): Participants randomized to the T&E Arm will initially receive 6 milligrams (mg) faricimab intravitreal (IVT) injections monthly (28d +/-7 days), with treatment intervals increased/extended, reduced, or maintained based on CST assessments, until week 100.
  Interventions: Drug: Faricimab
- Control/Usual Care Arm (Other): Participants in the control arm will receive 6 milligrams (mg) faricimab intravitreal (IVT) injections monthly (28d +/-7 days), for 6 treatments. Afterwards, participants will continue to receive 6mg faricimab IVT every 8 weeks until week 100.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered via intravitreal injection.

SUMMARY:
This study will assess a pragmatic, treat and extend regimen of faricimab against the standard of a fixed dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2).
3. Macular thickening secondary to DME (CI-DME) involving the center of the fovea on Optical Coherence Tomography - Central subfield thickness (CST) ≥ 325 μm on Spectralis at screening.***
4. Visual impairment due to DME, with best corrected visual acuity of 80 to 20 letters (Snellen VA 20/25 - 20/400).
5. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCT and fundus photographs.
6. Hemoglobin A1c must be <10% within 2 months prior to 1st study treatment.
7. Provide signed informed consent.

Exclusion Criteria:

1. Active or history of ocular inflammation or suspected/active ocular infection in either eye.
2. High-risk proliferative diabetic retinopathy in the study eye.**
3. Tractional retinal detachment, preretinal fibrosis or visually significant epiretinal membrane involving the macula.
4. Uncontrolled glaucoma (intraocular pressure >30 with or without medications).
5. Any intravitreal, periocular or implant corticosteroids within 26 weeks (6 months) before day 1 or any use of Iluvien implants.
6. Treatment with Panretinal photocoagulation (PRP) within 12 weeks before day 1.
7. Treatment with macular laser.
8. Any cataract surgery or any other intraocular surgery within 12 weeks before day 1.
9. Macular edema in study eye due to a cause other than DME.
10. If clinical exam and/or OCT and/or wide-field fluorescein angiography (WF-FA) suggest that (a) macular edema is considered to be related to ocular surgery such as cataract extraction or (b) if primary cause for macular edema is vitreoretinal interface abnormalities (e.g. a taut posterior hyaloid or epiretinal membrane).
11. Any ocular condition is present such that visual acuity loss would not improve from resolution of macular edema in opinion of the investigator (e.g. foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition)
12. Any history of ocular conditions that might affect macular edema (e.g. vein occlusion, idiopathic or infectious or non-infectious uveitis, ocular inflammatory disease, neovascular glaucoma etc.)
13. Women of child-bearing potential who are lactating, pregnant, or intending to become pregnant within the next 100 weeks.
14. Current or anticipated incarceration.
15. Terminal illness with expected survival less than 100 weeks.
16. Known hypersensitivity to faricimab or any of the excipients in the faricimab injection.
17. Currently enrolled in a study that does not permit co-enrollment.
18. Unable to obtain informed consent due to language or other operational barriers.
19. Anticipated problems, in the judgment of the site investigator, maintaining compliance with the protocol, including attending study visits, completing assessments or procedures.
20. Prior enrollment in this trial.
21. Other reason to exclude the patient, as approved by the sponsor and site investigator.
22. Previous treatment with anti-VEGF and:

    * <12 weeks prior to day 1 (washout period).*or,
    * Diagnosis of DME is > 2 years of enrollment or,
    * Do not have a demonstrated response to anti-VEGF treatment based on clinical discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity | Baseline to Week 100
  Change in best corrected visual acuity (3.9 letter non-inferiority margin)

SECONDARY OUTCOMES:
Decrease in Diabetic Retinopathy Severity Score | Baseline to Week 100
  A 2-step improvement in diabetic retinopathy severity score
Decrease in Diabetic Retinopathy Severity Score | Baseline to Week 100
  A 3-step improvement in diabetic retinopathy severity score
Change in Central Subfield Thickness | Baseline to Week 100
  Change in central subfield thickness on OCT
Change in Vision Related Quality of Life | Baseline to Week 100
  Change in vision-related quality of life (VFQ-25)
Change in Letters of Vision | Baseline to Week 100
  Gaining or losing ≥5, ≥10, or ≥15 letters of vision
Absence of Diabetic Macular Edema | Week 100
  Absence of diabetic macular edema in the study eye
Absence of Intraretinal Fluid (IRF) | Week 100
  Absence of intraretinal fluid (IRF) in the study eye
Dosing Interval | Week 100
  Dosing interval at week 100
Presence of Safety Outcomes | Baseline to Week 100
  Safety outcomes (ocular and systemic AEs and SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Varun Chaudhary, MD, FRCS(C), Principal Investigator — McMaster University
Locations (46):
- United States (11):
  - Retinal Consultants Medical Group Inc., Modesto, California
  - Vitreo-Retina Medical Group, Sacramento, California
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Eye Associates of Northeast Louisiana Dba Haik Humble Eye Center, West Monroe, Louisiana
  - Mississippi Retina Associates, Jackson, Mississippi
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Retina Consultants of Houston, dba Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retina Consultants of Houston, dba Retina Consultants of Texas, San Antonio, Texas
- Australia (16):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - Nexus Eyecare Blacktown, Blacktown, New South Wales
  - Eastern Suburbs Eye Specialists, Bondi Junction, New South Wales
  - Retina and Eye Consultants, Hurstville, New South Wales
  - Lane Cove Eye, Lane Cove, New South Wales
  - South West Retina, Liverpool, New South Wales
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - South Eastern Sydney Health, Sydney, New South Wales
  - Sydney Retina, Sydney, New South Wales
  - Queensland Eye Institute, Woolloongabba, Queensland
  - Adelaide Eye & Retina Centre, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - Lions Eye Institute Limited, Nedlands, Western Australia
- Canada (11):
  - Calgary Retina Consultants, Calgary, Alberta
  - Alberta Retina Consultants, Calgary, Alberta
  - Retina Surgical Associates, New Westminster, British Columbia
  - West Coast Retina, Vancouver, British Columbia
  - UBC Eye Centre, Vancouver General Hospital, Vancouver, British Columbia
  - The Research Institute of St. Joe's Hamilton, Hamilton, Ontario
  - St. Joseph's Healthcare London, London, Ontario
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Vitreous Retina Macula Specialists of Toronto, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- United Kingdom (8):
  - Bradford Royal Infirmary, Bradford, England
  - University Hospitals Bristol-Weston, Bristol, England
  - Frimley Health, Frimley, England
  - Liverpool University Hospitals, Liverpool, England
  - King's College Hospital, London, England
  - London North West University, London, England
  - Moorfields Eye Hospital, London, England
  - The Royal Wolverhampton, Wolverhampton, England